CLINICAL TRIAL: NCT05339503
Title: Comparison of Clinical Effectiveness of Hydrochloric Acid and Sodium Hypochlorite Used in Microabrasion Technique for the Treatment of Dental Fluorosis.
Brief Title: This is the Comparison of Clinical Effectiveness of Hydrochloric Acid-pumice Compound and Sodium Hypochlorite-pumice Compound Used in Microabrasion Technique for the Treatment of Dental Fluorosis. Change in Tooth Shade Was Checked Before and After the Procedure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Dental College (Other)
Responsible Party: Principal Investigator, HAREEM ABDUL SATTAR, Senior Registrar, Department of Operative Dentistry, Principal Investigator, Fatima Jinnah Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FatimaJDC
Record Dates: First submitted 2022-03-20; First posted 2022-04-21 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Dental Fluoroses
Keywords: Hydrochloric Acid; Sodium Hypochlorite; Dental Fluorosis; Microabrasion Technique
MeSH Terms: conditions — Fluorosis, Dental | interventions — Enamel Microabrasion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP A (HYDROCHLORIC ACID) (Experimental): Total 30 teeth in each group were included. Preoperatively shade was checked with VITA classical A1-D4® shade guide. The mixture (hydrochloric acid pumice compound) was applied 10 times or more during the same session. Total treatment time was around 30 minutes. Every patient received entire microabrasion treatment. At the end of the treatment, neutral sodium fluoride gel was applied. Then change in shade was checked again with VITA classical A1-D4® shade guide.
  Interventions: Other: enamel microabrasion
- GROUP B ( SODIUM HYPOCHLORITE) (Experimental): Total 30 teeth in each group were included. Preoperatively shade was checked with VITA classical A1-D4® shade guide.The mixture (sodium hypochlorite pumice compound) was applied 10 times or more during the same session. Total treatment time was around 30 minutes. Every patient received entire microabrasion treatment. At the end of the treatment, neutral sodium fluoride gel was applied. Then change in shade was checked again with VITA classical A1-D4® shade guide.
  .
  Interventions: Other: enamel microabrasion

INTERVENTIONS:
Other: enamel microabrasion — It is a non-restorative, conservative treatment that works both chemically and mechanically to remove up to 0.2 mm of affected enamel per application. Pumice either mixed with 18% hydrochloric acid or 5.25% sodium hypochlorite was used to remove fluorosis stains.

SUMMARY:
To compare the clinical effectiveness of hydrochloric acid-pumice compound and sodium hypochlorite-pumice compound in treating dental fluorosis using microabrasion technique.

DETAILED DESCRIPTION:
A Randomized Clinical Trial was taken Fatima Jinnah Dental College Hospital, Karachi, from 1st November 2019 To 30th April 2020. Total 30 teeth in each group were included. Preoperatively shade was checked. The mixture was applied 10 times or more during the same session. Total treatment time was around 30 minutes. Every patient received entire microabrasion treatment. At the end of the treatment, neutral sodium fluoride gel was applied. Then changes in shade were checked. Descriptive statistics were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 years .
* Permanent dentition assessed on clinical examination.
* Have at least four maxillary incisors with scores of 4 to 5, according to the Dean's Fluorosis Index.
* Have no caries or restoration on the teeth to be treated assessed clinically.

Exclusion Criteria:

* Poor oral dental and general health assessed on clinical examination.
* History of Smoking and any form of tobacco.
* Patients with periodontal disease assessed on clinical examination.
* Caries on anterior teeth assessed on clinical examination.
* Hypersensitive teeth assessed on clinical examination.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
HYDROCHLORIC ACID PUMICE COMPOUND | 30 minutes
  Tooth shade was recorded at the baseline with the help of VITA classical A1-D4® shade guide. The arrangement of the shades in the VITA classical family of shades is as follows: A1 - A4 (reddish-brownish), B1 - B4 (reddish-yellowish), C1 - C4 (greyish shades), D2 - D4 (reddish-grey).Determination of shade was done under daylight. Closest shade was selected from the shade tab. Effectiveness was marked positive if there was atleast one change in shade from the baseline just after the procedure to shade group from A1-D4. Effectiveness was marked negative if there is no change in shade from the baseline.
SODIUM HYPOCHLORITE PUMICE COMPOUND | 30 minutes
  Tooth shade was recorded at the baseline with the help of VITA classical A1-D4® shade guide. The arrangement of the shades in the VITA classical family of shades is as follows: A1 - A4 (reddish-brownish), B1 - B4 (reddish-yellowish), C1 - C4 (greyish shades), D2 - D4 (reddish-grey).Determination of shade was done under daylight. Closest shade was selected from the shade tab. Effectiveness was marked positive if there was atleast one change in shade from the baseline just after the procedure to shade group from A1-D4. Effectiveness was marked negative if there is no change in shade from the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: HAREEM A SATTAR, FCPS, Principal Investigator — Fatima Jinnah Dental College
Locations (1):
- Fatima Jinnah Dental College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
i will share the IPD once it will get published

REFERENCES:
- [Result] Nevarez-Rascon M, Molina-Frechero N, Adame E, Almeida E, Soto-Barreras U, Gaona E, Nevarez-Rascon A. Effectiveness of a microabrasion technique using 16% HCL with manual application on fluorotic teeth: A series of studies. World J Clin Cases. 2020 Feb 26;8(4):743-756. doi: 10.12998/wjcc.v8.i4.743. PMID 32149058
- [Result] Sheoran N, Garg S, Damle SG, Dhindsa A, Opal S, Gupta S. Esthetic management of developmental enamel opacities in young permanent maxillary incisors with two microabrasion techniques--a split mouth study. J Esthet Restor Dent. 2014 Sep-Oct;26(5):345-52. doi: 10.1111/jerd.12096. Epub 2014 Mar 4. PMID 24588784
- [Result] Gupta A, Dhingra R, Chaudhuri P, Gupta A. A comparison of various minimally invasive techniques for the removal of dental fluorosis stains in children. J Indian Soc Pedod Prev Dent. 2017 Jul-Sep;35(3):260-268. doi: 10.4103/JISPPD.JISPPD_138_16. PMID 28762354